CLINICAL TRIAL: NCT06947486
Title: COmparison of Physiological Dead Space Calculations Using EtCO₂ and P(A-a)O₂ in Mechanically Ventilated ICU Patients: A Prospective Observational Study
Brief Title: Correlation of EtCO₂- and P(A-a)O₂-Based Dead Space Calculations in Mechanically Ventilated ICU Patients
Acronym: CODE-EtA
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, A. Oguzhan KUCUK, MD, Assist Prof., Karadeniz Technical University
Other Study IDs: 2025/3
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Physiological Dead Space; Ventilation-Perfusion Mismatch; Mechanical Ventilation; Enghoff Correction
Keywords: Physiological Dead Space; EtCO₂; P(A-a)O₂ Gradient; Mechanical Ventilation; Volumetric Capnography; Ventilation-Perfusion Mismatch; Enghoff Modification; Kuwabara Equation; Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mechanically Ventilated ICU Patients: Adult patients (≥18 years old) admitted to a tertiary ICU and receiving invasive mechanical ventilation for at least 24 hours. Participants are prospectively monitored with capnographic and arterial blood gas measurements, and physiological dead space is calculated using both EtCO₂- and P(A-a)O₂-based methods. Patients are followed until ICU discharge or death.

SUMMARY:
This study aims to evaluate two different methods for calculating physiological dead space in adult patients undergoing invasive mechanical ventilation in the intensive care unit (ICU). Physiological dead space refers to the portion of air that is ventilated but does not participate in gas exchange due to impaired perfusion or ventilation-perfusion mismatch.

Traditionally, dead space is calculated using the end-tidal carbon dioxide (EtCO₂) method, which estimates the difference between arterial and exhaled CO₂ values. However, this method may be influenced by circulatory failure or abnormal CO₂ distribution. An alternative method using the alveolar-arterial oxygen gradient [P(A-a)O₂] has been proposed, as it may provide a more stable measurement under critical conditions by relying on oxygenation efficiency rather than CO₂ elimination.

In this prospective observational study, patients receiving mechanical ventilation in a tertiary ICU will be monitored. Physiological dead space will be calculated using both the EtCO₂-based method and the P(A-a)O₂-based method. Various respiratory and clinical parameters, including arterial blood gases, ventilator settings, and severity scores, will be recorded. The correlation between the two methods will be assessed, and their relationship with ICU mortality will be analyzed.

The results of this study may help determine whether the P(A-a)O₂ method can be used as a reliable alternative for estimating dead space in ICU patients and whether it has prognostic value in predicting patient outcomes.

DETAILED DESCRIPTION:
Physiological dead space (VD/VT) is a key parameter in evaluating the efficiency of gas exchange in mechanically ventilated patients. It represents the fraction of each breath that does not participate in effective alveolar ventilation due to perfusion defects, shunt physiology, or mismatched ventilation-perfusion (V/Q) ratios. An elevated dead space fraction has been associated with poor clinical outcomes, especially in patients with acute respiratory failure or circulatory impairment.

The most commonly used method for estimating dead space in the intensive care setting is based on the Enghoff modification of the Bohr equation:

VD/VT = (PaCO₂ - EtCO₂) / PaCO₂

This approach utilizes the arterial carbon dioxide pressure (PaCO₂) and end-tidal carbon dioxide pressure (EtCO₂) to estimate the proportion of ventilation that does not contribute to CO₂ elimination. However, it assumes a relatively homogenous V/Q distribution and may lose accuracy in the presence of increased shunt, circulatory shock, or CO₂ transport abnormalities.

To improve on these limitations, the present study also incorporates the alveolar-arterial oxygen gradient [P(A-a)O₂] as an alternative method for estimating physiological dead space. The gradient is calculated as:

P(A-a)O₂ = PAO₂ - PaO₂, where PAO₂ = FiO₂ × (Patm - PH₂O) - (PaCO₂ / R)

The dead space ratio can then be estimated by a similar structure:

VD/VT = (PAO₂ - PaO₂) / PAO₂

The P(A-a)O₂-based method may offer more robust estimations under critically ill conditions, particularly in cases with oxygenation defects or hemodynamic compromise, as it is less affected by variations in CO₂ distribution or metabolism.

In addition to Enghoff and oxygen-based approaches, this study also evaluates the Kuwabara modification, which adjusts for venous admixture and attempts to more accurately reflect the effective alveolar ventilation in the presence of shunt physiology. Kuwabara and Duncalf introduced a correction to the dead space formula to account for anatomical and functional shunts, reducing potential overestimation caused by disproportionate alveolar ventilation:

Corrected VD/VT = [(PaCO₂ - EtCO₂) / PaCO₂] × α

Where α represents a correction factor that adjusts for venous admixture and other circulatory influences.

This prospective observational study will include adult patients undergoing invasive mechanical ventilation in a tertiary ICU. Participants will be evaluated at multiple time points using volumetric capnography, arterial and venous blood gases, and ventilator-derived parameters. Physiological dead space will be calculated in parallel using:

Enghoff's method

P(A-a)O₂-based oxygenation gradients

Kuwabara correction for venous admixture

Daily clinical scores (SOFA, APACHE II), ventilator mechanics (PEEP, tidal volume, FiO₂, plateau pressure, driving pressure), and gas exchange variables (PaCO₂, PaO₂/FiO₂, VCO₂, VO₂) will also be recorded.

The study aims to assess:

The correlation between the EtCO₂- and P(A-a)O₂-based dead space methods

The influence of shunt and hemodynamic variables on dead space estimation

The prognostic relevance of each method in relation to ICU mortality

This study seeks to contribute to the optimization of dead space measurement in the ICU by evaluating alternative, potentially more reliable physiologic methods. It also aims to inform future clinical practice by identifying the most accurate and clinically useful dead space assessment tools in the context of severe critical illness.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission to the intensive care unit (ICU)
* Receiving invasive mechanical ventilation
* Expected ICU stay ≥ 24 hours
* Availability of both arterial blood gas and volumetric capnography measurements
* Central venous cathater for central venous blood analyses
* Informed consent obtained from legal representative

Exclusion Criteria:

* Refusal of participation by the patient or legal surrogate
* Hemoglobin < 7 g/dL
* PaCO₂ > 70 mmHg
* Lactate > 4 mmol/L
* Capillary refill time > 3 seconds
* Mean arterial pressure (MAP) < 65 mmHg
* Mottling score ≥ 2
* PaCO₂ - PcCO₂ gradient > 8 mmHg
* pH < 7.20
* Body temperature > 38°C
* BMI > 40 kg/m²
* VCO₂ > 4 mL/kg/min
* Technical limitations preventing accurate capnographic monitoring
* Patients who are extubated, transferred, or deceased within the first 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients (aged 18 years and older) who are admitted to a tertiary academic intensive care unit and require invasive mechanical ventilation for respiratory failure. Eligible patients must be expected to remain intubated for at least 24 hours and undergo both volumetric capnography and arterial blood gas monitoring. Participants are enrolled prospectively and consecutively based on predefined inclusion and exclusion criteria. Patients with circulatory shock, severe metabolic or respiratory derangements, or technical limitations interfering with capnographic measurement are excluded. The study represents a critically ill cohort commonly encountered in ICU practice.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2025-01-05 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Correlation between EtCO₂- and P(A-a)O₂-based dead space calculations | Within the first 72 hours of ICU admission
  Description: Pearson or Spearman correlation coefficient calculated between dead space values obtained from EtCO₂ (Enghoff modification) and P(A-a)O₂-based gradient methods in mechanically ventilated ICU patients.

SECONDARY OUTCOMES:
Association of each dead space method with ICU mortality | From ICU admission until ICU discharge or death
  Evaluation of whether EtCO₂- and P(A-a)O₂-derived dead space values are independently associated with ICU mortality.
Agreement between EtCO₂- and P(A-a)O₂-based dead space estimates | Within first 3 days of ICU stay
  Bland-Altman and bias analysis to evaluate agreement between the two measurement methods.
Relationship between dead space values and gas exchange/ perfusion variables | Daily for up to 72 hours
  Correlation between VD/VT and parameters such as PaO₂/FiO₂, lactate, MAP, and mottling score.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University Faculty of Medicine, Department of Chest Diseases, Intensive Care Unit, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and confidentiality considerations, and because no public data-sharing plan has been established for this study.